CLINICAL TRIAL: NCT05904470
Title: A Phase 2, Open-label Study to Assess the Safety and Efficacy of Bemnifosbuvir (BEM) and Ruzasvir (RZR) in Subjects With Chronic Hepatitis C Virus (HCV) Infection
Brief Title: A Phase 2, Safety and Efficacy of Bemnifosbuvir (BEM) and Ruzasvir (RZR) in Subjects With Chronic HCV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-01B-004
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Chronic Hepatitis C Virus; Hepatitis C, Chronic; Hepatitis C; Hepatic Cirrhosis; HCV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Liver Cirrhosis | interventions — AT-511; ruzasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Bemnifosbuvir and Ruzasvir (Experimental): Bemnifosbuvir (BEM; AT-527) Tablets
  Ruzasvir (RZR; AT-038) Capsules
  Interventions: Drug: Bemnifosbuvir; Drug: Ruzasvir

INTERVENTIONS:
Drug: Bemnifosbuvir — 550 mg administered orally once a day (QD) for 8 weeks
  Other Names: AT-527
Drug: Ruzasvir — 180 mg administered orally once a day (QD) for 8 weeks
  Other Names: AT-038

SUMMARY:
This is an open-label trial to evaluate safety and efficacy of treatment with BEM + RZR in subjects with chronic HCV infection.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Male or female subjects between ≥ 18 years of age (or the legal age of consent per local regulations) and ≤ 85 years of age
* Female subjects of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or to the use of an acceptable effective contraception
* Females must have a negative pregnancy test at Screening and at Day 1 prior to dosing
* Subjects must be direct-acting antiviral (DAA)-treatment-naïve, defined as never exposed to an approved or experimental DAA for HCV
* Documented medical history compatible with chronic HCV
* Liver disease staging assessment as follows:

  * Absence of cirrhosis (F0 to F3)
  * Compensated cirrhosis (F4)

Exclusion Criteria:

* Female subject is pregnant or breastfeeding
* Co-infected with hepatitis B virus (HBV; positive for hepatitis B surface antigen [HBsAg]) and/or human immunodeficiency virus (HIV)
* Abuse of alcohol and/or illicit drug use that could interfere with adherence to study requirements as judged by the investigator
* Prior exposure to any HCV DAA
* Use of other investigational drugs within 30 days of dosing or plans to enroll in another clinical trial of an investigational agent while participating in the present study
* Subject with known allergy to the study medications or any of their components
* History or signs of decompensated liver disease: ascites, variceal bleeding, hepatic encephalopathy, spontaneous bacterial peritonitis, or other clinical signs of portal hypertension or hepatic insufficiency
* Cirrhotic and has a Child-Pugh score >6, corresponding to a Child-Pugh Class B or C
* History of hepatocellular carcinoma (HCC) or findings suggestive of possible HCC
* Any other clinically significant medical condition that, in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2025-01-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- Atea Study Site, San Antonio, Texas, United States
- Brazil (12):
  - Atea Study Site, Manaus, Amazonas
  - Atea Study Site, Salvador, Estado de Bahia
  - Atea Study Site, Brasília, Federal District
  - Atea Study Site, Rio de Janeiro, Rio Do Janeiro
  - Atea Study Site, Porto Alegre, Rio Grande do Sul
  - Atea Study Site, Porto Velho, Rondônia
  - Atea Study Site, Boa Vista, Roraima
  - Atea Study Site, Botucatu, São Paulo
  - Atea Study Site, Ijuí, São Paulo
  - Atea Study Site, São José do Rio Preto, São Paulo
  - Atea Study Site, São Paulo, São Paulo
  - Atea Study Site, Sorocaba, São Paulo
- Canada (2):
  - Atea Study Site, Vancouver, British Columbia
  - Atea Study Site, Toronto, Ontario
- India (5):
  - Atea Study Site, Rajkot, Gujarat
  - Atea Study Site, Surat, Gujarat
  - Atea Study Site, Belagavi, Karnataka
  - Atea Study Site, Nagpur, Maharashtra
  - Atea Study Site, Kolkata, West Bengal
- Atea Study Site, Quatre Bornes, Mauritius
- Atea Study Site, Chisinau, Moldova
- Atea Study Site, Karachi, Pakistan
- Philippines (3):
  - Atea Study Site, Baguio City
  - Atea Study Site, Iloilo City
  - Atea Study Site, Mabalacat
- Romania (4):
  - Atea Study Site, Bucharest, BUC
  - Atea Study Site, Constanța, CON
  - Atea Study Site, Craiova, DOL
  - Atea Study Site, Bucharest
- South Africa (4):
  - Atea Study Site, Bloemfontein, Free State
  - Atea Study Site, Johannesburg, Gauteng
  - Atea Study Site, Randburg, Gauteng
  - Atea Study Site, Somerset West, Western Cap
- South Korea (4):
  - Atea Study Site, Seoul, Gyeonggi-do
  - Atea Study Site, Yangsan, Gyeongsangnam
  - Atea Study Site, Busan
  - Atea Study Site, Seoul
- Turkey (Türkiye) (5):
  - Atea Study Site, Adana
  - Atea Study Site, Ankara
  - Atea Study Site, Denizli
  - Atea Study Site, Izmir
  - Atea Study Site, Kayseri

RESULTS

PARTICIPANT FLOW:
Groups:
- BEM+RZR: Bemnifosbuvir (BEM; AT-527) 550 mg in combination with Ruzasvir (RZR; AT-038) 180 mg. Administered orally as two BEM tablets and two RZR capsules once a day (QD) for 8 weeks.
Period: Overall Study
Arm/Group | BEM+RZR
Started | 275
Completed | 255
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | BEM+RZR
Number analyzed (Participants) | 275
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (13.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131
  Male | 144
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 55
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 192
  More than one race | 3
  Unknown or Not Reported | 13
Genotype (GT) [Count of Participants; unit: Participants] — HCV genotypes are genetically distinct groups of HCV strains. Genotypes are classified based on differences in their nucleotide sequences and are used to categorize the virus into major types (which are numbered).
  Participants
    GT1 | 189
    GT2 | 7
    GT3 | 77
    GT4 | 2
Compensated Cirrhosis [Count of Participants; unit: Participants] | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Sustained Virologic Response at 12 Weeks Post-treatment (SVR12)
Description: SVR12 defined as plasma hepatitis C virus (HCV) RNA less than the lower limit of quantitation (<LLOQ) at 12 weeks post-treatment
Time Frame: Day 1 through 12 weeks after end of treatment
Population: The primary per-protocol analysis population included subjects who met all eligibility criteria, completed treatment (defined as being ≥90% compliant with the study drug regimen), had outcomes at post-treatment week 12, and had adequate study-drug exposure corroborated by pill counts and plasma drug levels adjudicated by an independent clinical pharmacologist.
Measure: Count of Participants; unit: Participants
Arm/Group | BEM+RZR
Number analyzed (Participants) | 215
Participants | 210

2. Secondary Outcome: Percentage of Subjects Experiencing Virologic Failure
Description: Virologic failure defined as a confirmed 1 log10 increase in HCV RNA from post-baseline nadir, or confirmed increase in HCV RNA ≥ LLOQ in any subject who achieved HCV RNA < LLOQ.
Time Frame: Day 1 through 12 weeks after end of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BEM+RZR
Number analyzed (Participants) | 215
Participants | 5

3. Secondary Outcome: Percentage of Subjects Achieving Sustained Virologic Response at 24 Weeks Post-treatment (SVR24)
Description: SVR24 defined as plasma HCV RNA less than the lower limit of quantitation (<LLOQ) at 24 weeks post-treatment
Time Frame: Day 1 through 24 weeks after end of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BEM+RZR
Number analyzed (Participants) | 211
Participants | 206

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected through 4 weeks post-treatment and serious adverse events were collected through 24 weeks post-treatment.
Arm/Group | BEM+RZR
All-Cause Mortality (participants affected / at risk) | 5/275
Serious Adverse Events (participants affected / at risk) | 19/275
Other Adverse Events (participants affected / at risk) | 64/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BEM+RZR (N=275)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Behaviour disorder (Psychiatric disorders) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Death (General disorders) | 1 (1) — cause unknown
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BEM+RZR (N=275)
Headache (Nervous system disorders) | 24
Nausea (Gastrointestinal disorders) | 22
Dyspepsia (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 12
Pyrexia (General disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 10
Fatigue (General disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 6

LIMITATIONS AND CAVEATS:
This was a single arm study. Results will need to be confirmed in larger, controlled randomized trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator may publish or present results pertaining to the PI's activities after the first publication of the multicentre clinical trial results. Publication or presentation of data from individual study centers is subject to prior review by the Sponsor. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT05904470/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT05904470/SAP_001.pdf